CLINICAL TRIAL: NCT06579209
Title: NAD+ Oral Supplement Pilot Intervention in Adult Females
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rhode Island (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2087241-4; P20GM103430 (NIH)
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Cognitive Change; Inflammation; Neurodegenerative Diseases
MeSH Terms: conditions — Inflammation; Neurodegenerative Diseases | interventions — NAD

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pre-testing prior to intervention (No Intervention): Prior to receiving the supplement, either Nicotinamide adenine dinucleotide or the placebo, participants will undergo cognitive testing and a blood draw.
- Post-testing after intervention (No Intervention): After receiving the supplement, either Nicotinamide adenine dinucleotide or the placebo, participants will undergo cognitive testing and a blood draw.
- Intervention (Experimental): For four weeks, the participant will consume an oral supplement, either Nicotinamide adenine dinucleotide or a placebo.
  Interventions: Dietary Supplement: Nicotinamide adenine dinucleotide

INTERVENTIONS:
Dietary Supplement: Nicotinamide adenine dinucleotide — Participants will take a supplement for four weeks. The supplement will either be Nicotinamide adenine dinucleotide or a placebo
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to learn if Nicotinamide adenine dinucleotide (NAD+) can influence cognition and biomarkers in healthy, cognitively intact women who identify as Latina and are between the ages of 40-80. The main questions it aims to answer are:

Will executive function change in response to NAD+? Will inflammatory markers and serum indicators of neurodegeneration change in response to NAD+? Researchers will compare individuals receiving the NAD+ to see if the results differ from those receiving the placebo.

Participants will:

Complete an online questionnaire, Visit the lab for computerized cognitive testing and a blood draw, Take NAD+ or a placebo every day for 4 weeks, Visit the lab for computerized cognitive testing and a blood draw

ELIGIBILITY:
Inclusion Criteria:

* Identify as Latina, have three or more adverse childhood experiences, and a BMI of 18.5 or above

Exclusion Criteria:

* Those who are taking hormone medication, pregnant or breastfeeding

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-reported biological sex
Enrollment: 50 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Neurocognition | four weeks
  NIH Toolkit Cognition Battery, Automated Neuropsychological Assessment Metrics
Neurodegenerative disease panel | four weeks
  BDNF, Cathespin D, MPO, PAI-1 (total), PDGF-AA, PDGF-AB/BB, RANTES, slCAM-1, sNCAM, sVCAM-1
Markers of systemic inflammation | four weeks
  GM-CSF, IFNγ, IL-1β, IL-2, IL-4, IL-5, IL-6, IL-8, IL-10, IL-12p70, IL-13, IL-17A, IL-23, TNFα

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Rhode Island, Kingston, Rhode Island
  - Independence Square, University of Rhode Island, Pawtucket, Rhode Island

IPD SHARING:
Plan to Share IPD: No